CLINICAL TRIAL: NCT00833469
Title: Escitalopram for the Treatment of Postpartum Depression
Brief Title: Escitalopram (Lexapro) for the Treatment of Postpartum Depression
Acronym: LexaproPPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Marlene P. Freeman, MD, Clinical Director, Center for Women's Mental Health, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-P-001509
Record Dates: First submitted 2009-01-29; First posted 2009-02-02 (Estimated); Results first posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Postpartum Depression
Keywords: women; postpartum depression; anxiety
MeSH Terms: conditions — Depression, Postpartum; Anxiety Disorders | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Escitalopram (Experimental): Flexible dose escitalopram 10mg
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Once daily by mouth
  Other Names: Lexapro

SUMMARY:
The purpose of this study is to determine whether women with postpartum major depressive disorder (MDD) will experience a significant decrease in depressive symptoms from baseline over an eight-week treatment intervention with escitalopram (Lexapro). Also, to determine whether women with postpartum MDD will experience a significant decrease in anxiety symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18 to 45 years old
* Subjects must meet criteria for a major depressive episode with symptoms developing within three month of live childbirth
* Subjects must present within six months of childbirth
* MADRS score >15
* BAI score >10
* Subjects will be able to be treated on an outpatient basis
* Subjects will be able to provide written informed consent

Exclusion Criteria:

* Subjects who have taken any psychotropic medication, including antidepressants and anti-anxiety medication, within the past two weeks (with the exception of non-benzodiazepine medications used for sleep, including trazodone, zolpidem, eszopiclone, etc)
* Suicidal ideation with active plan or intent, as determined by the investigator
* Presence of psychotic symptoms or homicidal ideation
* History of mania or hypomania
* Pregnant or breastfeeding
* Presence of chronic depression or dysthymia, or chronic or treatment resistant anxiety disorders, as determined by investigator
* Active alcohol/substance abuse currently or within the past year
* Abnormal TSH, severe anemia, or uncontrolled hypertension

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2009-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marlene P Freeman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: Center for Women's Mental Health Online Resource — http://www.womensmentalhealth.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Seven subjects were enrolled in this study. Prior to receiving treatment, two subjects were found to be ineligible per protocol eligibility requirements.
Groups:
- Escitalopram: Flexible dose escitalopram 10mg once daily by mouth (maximum of 20mg, minimum of 5mg, per the investigator's discretion).
Period: Overall Study
Arm/Group | Escitalopram
Started | 5
Completed | 3
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Of the 7 subjects consented, 5 were eligible to initiate study intervention. Out of these 5, 1 subject dropped prior to V1 and no baseline information is available for her.
Arm/Group | Escitalopram
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinician-rated Montgomery-Asberg Depression Rating Scale (MADRS)
Description: The Montgomery-Åsberg Depression Rating Scale is a widely used 10-item clinician-rated scale that describes the severity of depressive symptoms (range 0-60, higher score indicates greater symptom burden).
Time Frame: 8 weeks
Population: Of 7 subjects consented, 5 were eligible after V1. Before V2, 1 subject dropped and 1 was LTF. Three subjects completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escitalopram
Number analyzed (Participants) | 3
units on a scale | -21.33 (11.24)

2. Secondary Outcome: Change in Edinburgh Postnatal Depression Scale (EPDS)
Description: The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self-report used to measure postpartum depression (range 0-30, higher score indicates greater symptom burden). A score of >9 is indicative of perinatal major depression.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escitalopram
Number analyzed (Participants) | 3
units on a scale | -19.33 (2.52)

3. Secondary Outcome: Change in Beck Anxiety Inventory (BAI)
Description: Beck Anxiety Inventory (BAI): The BAI is a 21-item self-report questionnaire measuring typical symptoms of anxiety during the past week (range 0-63, higher score indicates greater anxiety).
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escitalopram
Number analyzed (Participants) | 3
units on a scale | -15.00 (9.85)

ADVERSE EVENTS:
Time Frame: 32 months
Arm/Group | Escitalopram
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Escitalopram (N=3)
Nausea (Gastrointestinal disorders) | 2
Decreased sleep (Nervous system disorders) | 1
Jaw tightness (Musculoskeletal and connective tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1

LIMITATIONS AND CAVEATS:
We recruited only 7 patients out of a projected 20. Patients were not referred because they were breastfeeding or preferred to receive treatment from their primary care doctor. We also suspect that many women with PPD do not seek treatment at all.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No